CLINICAL TRIAL: NCT03432988
Title: Impact of Nurses´ Solution-focused Communication on the Fluid Adherence of Adult Patients on Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, María del Carmen Neipp, PhD, Universidad Miguel Hernandez de Elche
Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: UMH-SFNursing
Record Dates: First submitted 2018-02-06; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Renal Dialysis
Keywords: Nursing Solution-Focused; hemodialysis; Psychosocial intervention; Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nurses in the hemodialysis service (Experimental): Nursing Solution-Focused: Two two-hour training modules were designed by two recognized solution-focused therapy experts. In each module, participants watched videos that illustrated solution-focused communication on fluid adherence, and practiced the skills in role-plays.
  Interventions: Behavioral: Nursing Solution-Focused

INTERVENTIONS:
Behavioral: Nursing Solution-Focused — Two two-hour training modules were designed. In each module, participants watched videos that illustrated solution-focused communication on fluid adherence, and practiced the skills in role-plays. Solution-focused communication on IDWG. In the case of IDWG improvement, nurses were trained to congratulate the patient and then to explore in detail, from a stance of curiosity, how s/he had accomplished the weight reduction. Nurses were trained to invite patients to share specific behavioral details, to describe their own behavior from the perspective of significant family members and also to compliment patients on their accomplishments and to invite them to keep track of anything else they might find useful to control fluid intake over the next days.

SUMMARY:
Aim: To test the hypothesis that fluid adherence in patients on hemodialysis can be improved through nurses´ solution-focused communication with patients on issues of adherence.

Design: Single-group quasi-experimental study. Method: A one-month baseline of inter-dialytic weight gain was taken for a group of 36 adult patients in a hospital hemodialysis unit. Then, the nurses of the unit received an 5-hour training in solution-focused communication on issues of fluid adherence and applied it with the patients of the sample. Inter-dialytic weight gains (IDWG) were measured during another month. Six months after the training, IDWG was again measured during one month.

DETAILED DESCRIPTION:
Design A single-group quasi-experimental design was carried out. The IDWG was the dependent variable, expressed as the weight gain in kilograms between dialysis sessions. A base-line was established by taking IDWG data for one month; after the nurses training, IDWG data were taken for another month. Follow-up was carried out six months later.

Methods

Participants 36 patients of a hemodialysis unit in a public hospital were invited to participate in the study. All accepted and gave written informed consent. Nurses were two women (39 and 37 years old) and one man (30 years old).

The intervention Training. Two two-hour training modules were designed by two recognized solution-focused therapy experts. In each module, participants watched videos that illustrated solution-focused communication on fluid adherence, and practiced the skills in role-plays.

Solution-focused communication on IDWG. In the case of IDWG improvement, nurses were trained to congratulate the patient and then to explore in detail, from a stance of curiosity, how nurses had accomplished the weight reduction. Nurses were trained to invite patients to share specific behavioral details and also to describe their own behavior from the perspective of significant family members. Nurses were also taught to compliment patients on their accomplishments and to invite them to keep track of anything else they might find useful to control fluid intake over the next days.

In the case of IDWG worsening, nurses were encouraged to validate patients´ difficulties and empathize with their predicament.

A repeated measure analysis of variance (ANOVA) and Student's t were used to analyze the changes in patient's IDWG over time.

ELIGIBILITY:
Inclusion Criteria:

* 0

Exclusion Criteria:

* 0

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
ANOVA | Three months
  Analysis of Variance

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pastor, Study Chair — Universidad Miguel Hernández de Elche
Locations (1):
- María del Carmen Neipp, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Starting one month after publication
Access Criteria: Researcher should write an email to the principal investigator, telling the reasons for asking for the data

REFERENCES:
- [Background] Baines LS, Jindal RM. Non-compliance in patients receiving haemodialysis: an in-depth review. Nephron. 2000 May;85(1):1-7. doi: 10.1159/000045622. No abstract available. PMID 10773748
- [Background] Idier L, Untas A, Koleck M, Chauveau P, Rascle N. Assessment and effects of Therapeutic Patient Education for patients in hemodialysis: a systematic review. Int J Nurs Stud. 2011 Dec;48(12):1570-86. doi: 10.1016/j.ijnurstu.2011.08.006. Epub 2011 Sep 14. PMID 21924423
- [Background] Kugler C, Maeding I, Russell CL. Non-adherence in patients on chronic hemodialysis: an international comparison study. J Nephrol. 2011 May-Jun;24(3):366-75. doi: 10.5301/JN.2010.5823. PMID 20954134
- [Background] McAllister M. Doing practice differently: solution-focused nursing. J Adv Nurs. 2003 Mar;41(6):528-35. doi: 10.1046/j.1365-2648.2003.02564.x. PMID 12622862
- [Background] McGee D, Del Vento A, Bavelas JB. An interactional model of questions as therapeutic interventions. J Marital Fam Ther. 2005 Oct;31(4):371-84. doi: 10.1111/j.1752-0606.2005.tb01577.x. No abstract available. PMID 16294686
- [Background] Morgan L. A decade review: methods to improve adherence to the treatment regimen among hemodialysis patients. Nephrol Nurs J. 2000 Jun;27(3):299-304. PMID 11249328
- [Background] Matteson ML, Russell C. Interventions to improve hemodialysis adherence: a systematic review of randomized-controlled trials. Hemodial Int. 2010 Oct;14(4):370-82. doi: 10.1111/j.1542-4758.2010.00462.x. Epub 2010 Aug 27. PMID 20796047
- [Background] Bowles N, Mackintosh C, Torn A. Nurses' communication skills: an evaluation of the impact of solution-focused communication training. J Adv Nurs. 2001 Nov;36(3):347-54. doi: 10.1046/j.1365-2648.2001.01979.x. PMID 11686749
- [Derived] Beyebach M, Neipp MDC, Garcia-Moreno M, Gonzalez-Sanchez I. IMPACT of nurses' solution-focused communication on the fluid adherence of adult patients on haemodialysis. J Adv Nurs. 2018 Nov;74(11):2654-2657. doi: 10.1111/jan.13792. Epub 2018 Aug 19. PMID 29992599